CLINICAL TRIAL: NCT06069713
Title: The Impact of Cannabidiol (CBD) Health Claims at Point-of-Sale on Consumer Perceptions and Behavior: Online Survey
Brief Title: Consumer Perceptions of Cannabidiol (CBD) Health Claims
Acronym: CBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of North Carolina, Chapel Hill (Other); Public Health Law Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00094734; 1R01DA051542 (NIH)
Record Dates: First submitted 2023-09-21; First posted 2023-10-06 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2023-06

CONDITIONS: Perceptions
Keywords: CBD; Cannabidiol; Marketing; Health claims

STUDY DESIGN:
Intervention Model Description: Conduct a cross-sectional online survey with a nationally representative probability-based sample of adults, ages 18-65 to assess consumer perceptions of 55 documented advertisements about CBD. Participants will be randomly assigned to 1 of 11 panels that each contain 5 advertisements about CBD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perception of Ads (Experimental): Each panel will consist of 5 different advertisements for CBD. With 11 panels and 5 images each, there are a total of 55 images that will be viewed by the participants. Participants will view an image, one at a time, and answer questions about their perceptions of the advertisement.
  Interventions: Behavioral: CBD advertisements

INTERVENTIONS:
Behavioral: CBD advertisements — Participants will view the 5 images of CBD advertisements in their assigned panel and answer questions about their perceptions of the advertisement.
  Other Names: images of CBD advertisements

SUMMARY:
Over 46 million US adults report use of cannabidiol (CBD), primarily to treat medical ailments. The growing CBD market spans the range of products that the US Food and Drug Administration (FDA) regulates including drugs, dietary supplements, food/beverages and cosmetics. CBD cannot be marketed as having therapeutic benefits (without FDA's approval), be false or misleading to consumers, or convey the products are approved or endorsed by the FDA. In addition, CBD cannot be marketed as a food additive or dietary supplement since it is an active ingredient in an approved drug, Epidiolex. Despite this, CBD products have been illicitly advertised to consumers with these claims including unsubstantiated health claims that promote benefits including curing cancer and preventing Alzheimer's disease. These types of claims may reduce perceptions of harm and increase perceived benefits of use. This study aims to evaluate how consumers perceive real-world CBD advertisements. To that end, we will implement an online survey and randomize adult participants (ages 18-65) to see various advertisements made about CBD to determine if they interpret advertisements as making health claims that are currently prohibited by the FDA.

DETAILED DESCRIPTION:
Cannabidiol (CBD) products have rapidly gained popularity, spanning the retail market with a range of products that the US Food and Drug Administration (FDA) regulates including drugs, dietary supplements, food/beverages and cosmetics. The FDA mandates that CBD cannot be marketed as having therapeutic benefits (without FDA's approval), be false or misleading to consumers, or convey the products are approved or endorsed by the FDA. In addition, CBD cannot be marketed as a food additive or dietary supplement since it is an active ingredient in an approved drug, Epidiolex. Despite this, CBD products have been unlawfully advertised to consumers with these claims including unsubstantiated health claims that promote benefits including curing cancer and preventing Alzheimer's disease and providing chronic pain relief. This project, focused on informing regulatory actions for CBD, aims to evaluate consumer perceptions of real-world health claims documented in brick and mortar CBD retailers in three US states.

Setting: The survey will be a single online experiment with one survey. The survey will last approximately 20 minutes.

Recruitment: Adult CBD and non-CBD users, ages 18-65, will be recruited through NORC, an online survey panel company. Interested prospective participants will complete a screening questionnaire to determine their eligibility. If eligible, NORC will invite them to enroll in the study. Approximately 3525 participants will complete the study.

Informed consent: Participants will provide online consent prior to the main survey, after determining eligibility.

Randomization: After providing informed consent, participants will be randomly assigned to one of eleven panels. Participants will have an equal chance of being randomized to any of the eleven panels. Each panel will view 5 advertisements about CBD that was documented in a CBD retailer in the US.

Assessment: Participants in the study will complete one survey that will take approximately 20 minutes. During the survey, participants will view 5 advertisements about CBD. Participants will be randomized to 1 of 11 panels, each containing 5 different advertisements. Within each panel, participants will be randomized to the order of the images they see and will be asked a series of questions after each advertisement to determine the appeal CBD and if they perceive the ad to be making health claims that are prohibited by the US FDA. After viewing all 5 ads in their assigned panel, participants will complete measures assessing outcome expectancies of CBD use, perceived benefits of daily CBD use, and willingness to try CBD (non-users only).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* US Residents
* Satisfies one of the following categories:

  1. Current CBD users
  2. Ever CBD users
  3. Non-CBD users
* Members of the AmeriSpeak™ panel

Exclusion Criteria:

* Non-English speakers
* Younger than 18 or older than 65
* Not US residents
* Not members of the AmeriSpeak™ panel

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3504 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Wagoner, Dr.PH, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 people were consented but dropped out of the study prior to being assigned a panel. 428 people were excluded from analysis due to poor data quality: The excluded ppts did not meet sufficient completion criteria. Participants must have met both of the following criteria to be included in the study: 1) at least 75% of the outcome variables answered (not skipped) and 2) survey completion time of > 5min
Groups:
- Panel 1; Panel 2; Panel 3; Panel 4; Panel 5; Panel 6; Panel 7; Panel 8; Panel 9; Panel 10; Panel 11: This panel consists of 5 photos that were found in CBD retail assessments. Photos were coded as at least one of six FDA prohibited claim types or contained product descriptors that may be potentially misleading to consumers. Photos did not differ substantially between panels and panels were only used to reduce participant burden, as 55 photos were to be included in the survey
Period: Overall Study
Arm/Group | Panel 1 | Panel 2 | Panel 3 | Panel 4 | Panel 5 | Panel 6 | Panel 7 | Panel 8 | Panel 9 | Panel 10 | Panel 11
Started | 307 | 311 | 307 | 305 | 334 | 319 | 292 | 301 | 346 | 354 | 328
Completed | 262 | 281 | 276 | 262 | 289 | 280 | 253 | 266 | 302 | 312 | 293
Not Completed | 45 | 30 | 31 | 43 | 45 | 39 | 39 | 35 | 44 | 42 | 35

BASELINE CHARACTERISTICS:
Population: 21 people were consented but dropped out of the study prior to being assigned a panel. 428 people were excluded from analysis due to poor data quality: The excluded ppts did not meet sufficient completion criteria. Participants must have met both of the following criteria to be included in the study: 1) at least 75% of the outcome variables answered (not skipped) and 2) survey completion time of > 5min
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel 1 | Panel 2 | Panel 3 | Panel 4 | Panel 5 | Panel 6 | Panel 7 | Panel 8 | Panel 9 | Panel 10 | Panel 11 | Total
Number analyzed (Participants) | 262 | 281 | 276 | 262 | 289 | 280 | 253 | 266 | 302 | 312 | 293 | 3076
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (13.1) | 43.8 (12.8) | 43.5 (13.8) | 43.9 (13.7) | 43.9 (14.3) | 43.2 (13.1) | 43.7 (13.8) | 43.9 (13.3) | 44.0 (13.4) | 43.8 (14.0) | 43.1 (13.5) | 43.6 (13.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Current Gender Male | 121 | 119 | 121 | 113 | 121 | 131 | 105 | 119 | 133 | 142 | 128 | 1353
  Current Gender Female | 132 | 156 | 146 | 142 | 159 | 143 | 142 | 140 | 157 | 159 | 156 | 1632
  Current Gender Transgender | 1 | 2 | 3 | 2 | 0 | 1 | 1 | 2 | 3 | 2 | 1 | 18
  None of the Above Genders | 1 | 0 | 0 | 1 | 3 | 1 | 2 | 4 | 3 | 2 | 2 | 19
  Did not answer | 7 | 4 | 6 | 4 | 6 | 4 | 3 | 1 | 6 | 7 | 6 | 54
  Sex assigned at birth Male | 122 | 119 | 124 | 114 | 125 | 131 | 108 | 122 | 134 | 145 | 128 | 1372
  Sex assigned at birth Female | 134 | 157 | 146 | 143 | 157 | 144 | 142 | 142 | 160 | 160 | 155 | 1640
  Sex assigned at birth Did not answer | 6 | 5 | 6 | 5 | 7 | 5 | 3 | 2 | 8 | 7 | 10 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 21 people were consented but dropped out of the study prior to being assigned a panel. 428 people were excluded from analysis due to poor data quality: The excluded ppts did not meet sufficient completion criteria. Participants must have met both of the following criteria to be included in the study: 1) at least 75% of the outcome variables answered (not skipped) and 2) survey completion time of > 5min
  Participants
    Hispanic or Latino | 218 | 247 | 227 | 233 | 238 | 254 | 217 | 230 | 263 | 274 | 259 | 2660
    Not Hispanic or Latino | 44 | 34 | 49 | 29 | 51 | 26 | 36 | 36 | 39 | 38 | 34 | 416
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 2 | 0 | 0 | 3 | 1 | 2 | 2 | 4 | 0 | 17
  Asian | 11 | 15 | 6 | 15 | 8 | 7 | 7 | 10 | 14 | 15 | 10 | 118
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 9
  Black or African American | 35 | 26 | 34 | 31 | 46 | 37 | 33 | 39 | 40 | 48 | 45 | 414
  White | 195 | 213 | 199 | 195 | 202 | 214 | 187 | 190 | 220 | 216 | 211 | 2242
  More than one race | 8 | 13 | 15 | 13 | 20 | 10 | 15 | 16 | 12 | 12 | 16 | 150
  Unknown or Not Reported | 11 | 10 | 19 | 8 | 13 | 8 | 10 | 9 | 12 | 15 | 11 | 126
Education Level [Count of Participants; unit: Participants]
  Less than High School | 15 | 13 | 26 | 17 | 23 | 20 | 13 | 15 | 13 | 19 | 24 | 198
  HS graduate or equivalent | 43 | 56 | 48 | 41 | 53 | 49 | 33 | 34 | 55 | 48 | 54 | 514
  Vocational/tech school/some college/associates | 98 | 87 | 99 | 104 | 115 | 109 | 89 | 94 | 115 | 119 | 97 | 1126
  Bachelor's Degree | 70 | 72 | 57 | 63 | 55 | 66 | 74 | 75 | 65 | 89 | 77 | 763
  Post grad study/professional degree | 36 | 53 | 46 | 37 | 43 | 36 | 44 | 48 | 54 | 37 | 41 | 475
SES [Count of Participants; unit: Participants]
  Less than $10,000 | 9 | 9 | 19 | 9 | 17 | 14 | 6 | 16 | 12 | 18 | 15 | 144
  $10,000 to less than $25,000 | 20 | 42 | 32 | 32 | 27 | 33 | 25 | 33 | 34 | 30 | 35 | 343
  $25,000 to less than $50,000 | 44 | 48 | 51 | 60 | 64 | 61 | 52 | 49 | 70 | 67 | 64 | 630
  $50,000 to less than $75,000 | 59 | 54 | 60 | 47 | 56 | 59 | 40 | 46 | 50 | 50 | 52 | 573
  $75,000 to less than $100,000 | 37 | 43 | 33 | 31 | 52 | 40 | 47 | 39 | 31 | 43 | 42 | 438
  More than $100,000 | 93 | 85 | 81 | 83 | 73 | 73 | 83 | 83 | 105 | 104 | 85 | 948
State Cannabis policy [Count of Participants; unit: Participants]
  Medical and Recreational states | 151 | 149 | 135 | 145 | 163 | 155 | 143 | 143 | 161 | 172 | 169 | 1686
  Medical only states | 48 | 62 | 71 | 54 | 53 | 57 | 54 | 60 | 62 | 62 | 56 | 639
  CBD/Low THC states | 54 | 61 | 62 | 58 | 65 | 59 | 52 | 53 | 72 | 68 | 59 | 663
  No cannabis access states | 9 | 9 | 8 | 5 | 8 | 9 | 4 | 10 | 7 | 10 | 9 | 88

OUTCOME MEASURES:

1. Primary Outcome: Perceived Claim Scores
Description: The primary outcome is consumer perception of the claims in the ads (n=55) and whether perceptions of prohibited claims vary by CBD use status. After viewing each of the 5 assigned ads participants will respond to six items that assess their perception of the prohibited claims made in the ads, including 1) drug effect 2) FDA approved/ endorsed 3) dietary supplement 4) food additive 5) false/misleading (scientific) and 6) false/misleading (targeting youth). The Study Team will use a 5-point response scale, (1) Not at all to (5) Extremely to assess perception of each prohibited claim type. For each use status group, the Study Team will report the overall mean score (all ads together) for each claim type to indicate if perception of prohibited claims differed by use status.
Time Frame: Minute 15
Population: participants were pre-specified to be reported "per CBD user status"
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Current CBD Users: Participants who have used CBD in the last month
- Ever CBD Users: Participants who have used CBD before, but not in the last month
- Non CBD Users: Participants who have never used CBD
Arm/Group | Current CBD Users | Ever CBD Users | Non CBD Users
Number analyzed (Participants) | 1008 | 1053 | 1015
score on a scale
  Drug Effect | 2.96 (0.02) | 2.81 (0.02) | 2.71 (0.03)
  FDA | 2.03 (0.03) | 1.76 (0.02) | 1.64 (0.02)
  Dietary Supplement | 2.44 (0.02) | 2.23 (0.02) | 2.18 (0.02)
  Food Additive | 2.32 (0.03) | 2.06 (0.02) | 2.00 (0.02)
  False and Misleading (Science) | 2.57 (0.03) | 2.27 (0.02) | 2.11 (0.02)
  False and Misleading (Youth) | 2.68 (0.02) | 2.55 (0.02) | 2.57 (0.02)

2. Secondary Outcome: Perceived Product Safety Scores
Description: For each ad that the participant views (n=5), the Participant will respond to a one-item measure that assesses the extent to which the participant perceives that CBD is safe to consume. Response options are on a 1 to 5 scale, with higher scores representing more perceived safety (i.e. 1- Not at all safe to 5- Extremely safe). For each use status group, the Study Team will report the mean score of perceived safety to indicate if the perceived safety of CBD in the advertisements differed by use status.
Time Frame: Minute 15
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Non-CBD Users: Participants who have never used CBD
Arm/Group | Current CBD Users | Ever CBD Users | Non-CBD Users
Number analyzed (Participants) | 1008 | 1053 | 1015
score on a scale | 3.34 (0.02) | 3.11 (0.02) | 2.92 (0.03)

3. Secondary Outcome: Appeal Scores
Description: For each ad that the participant views (n=5), the Participant will respond to a one-item measure to assess the extent to which the ad makes CBD appealing to them. Response options are on a 1 to 5 scale, with higher scores representing more appeal (i.e. 1- Not at all appealing to 5- Extremely appealing). For each use status group, the Study Team will report the mean score of appeal to indicate if the appeal of CBD in the advertisements differed by use status.
Time Frame: Minute 15
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Current CBD Users | Ever CBD Users | Non-CBD Users
Number analyzed (Participants) | 1008 | 1053 | 1015
score on a scale | 2.82 (0.02) | 2.42 (0.02) | 1.81 (0.02)

4. Other Pre Specified Outcome: Outcome Expectancies Scores
Description: Ten items will measure participants' perceptions about the possible effects of CBD. Response items are on a 1 to 5 scale, with higher scores representing more agreement with the stated effect (i.e. 1- Strongly disagree to 5- Strongly agree).
Time Frame: Minute 15
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Perceived Benefit Scores
Description: Seventeen items will measure participants' perceived benefits of daily CBD use to treat various medical conditions. Response items are on a 1 to 4 scale (1-Worsen the condition; 2- No effect on the condition; 3-Improve the condition; 4- I don't know)
Time Frame: Minute 15
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Willingness to Try Cannabidiol (CBD) (Non-CBD Users Only) Scores
Description: One item will be used to measure non-user's willingness to try CBD. Response items are on a 1 to 5 scale, with higher scores representing more likelihood to try CBD (i.e. 1- Extremely Unlikely to 5- Extremely Likely)
Time Frame: Minute 15
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Week 5
Groups:
- Ever CBD Users: Participants who have used CBD but not in the past month
Arm/Group | Current CBD Users | Ever CBD Users | Non CBD Users
All-Cause Mortality (participants affected / at risk) | 0/1008 | 0/1053 | 0/1015
Serious Adverse Events (participants affected / at risk) | 0/1008 | 0/1053 | 0/1015
Other Adverse Events (participants affected / at risk) | 0/1008 | 0/1053 | 0/1015

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT06069713/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT06069713/ICF_000.pdf